CLINICAL TRIAL: NCT01762189
Title: Multicenter Prospective Study on the Incidence and Risk Factors of Neonatal Hyperbilirubinemia in Term and Late-preterm Chinese Infants
Brief Title: The Incidence and Risk Factors of Neonatal Hyperbilirubinemia in Term and Late-preterm Chinese Infants
Status: Completed | Type: Observational
Sponsor: Nanjing Medical University (Other)
Collaborators: Children's Hospital of Fudan University (Other); Nanjing Maternity and Child Health Care Hospital (Other); Jinlin Provincial Maternal and Child Health Hospital (Unknown); Peking University Third Hospital (Other); Inner Mongolia Maternal and Child Health Care Hospital (Other); Shanxi Provincial Maternity and Children's Hospital (Other); Obstetrics & Gynecology Hospital of Fudan University (Other); Guangdong Women and Children Hospital (Other); Guangxi Maternal and Child Health Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); First Affiliated Hospital of Xinjiang Medical University (Other); First Affiliated Hospital of Harbin Medical University (Other); Sichuan Provincial People's Hospital (Other); Guiyang Maternity and Child Health Care Hospital (Other)
Responsible Party: Principal Investigator, Zhangbin Yu, Principal Investigator, Nanjing Medical University
Other Study IDs: NMU-FY2012-319
Record Dates: First submitted 2013-01-02; First posted 2013-01-07 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Hyperbilirubinemia, Neonatal
Keywords: Hyperbilirubinemia; Neonatal; Incidence; Risk factors
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia | interventions — Phototherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Phototherapy — The decision to use phototherapy conformed to the hour-specific threshold value for phototherapy presented by the American Academy of Pediatrics guidelines and was not at the discretion of the investigators.

SUMMARY:
Thirteen hospitals in China will participate in the study, which aims to provide data on serum bilirubin levels in the first 168 hr after birth in term and late-preterm neonates, and estimate the incidence of severe neonatal hyperbilirubinemia and the underlying causes.

We hypothesize that the study can be value in identifying and implementing strategies for risk reduction.

DETAILED DESCRIPTION:
Neonatal hyperbilirubinemia resulting in clinical jaundice is a common problem among infants, particularly during the first weeks of life.

Information about the incidence and risk factors of neonatal jaundice is not available from China where is one of the highest countries of the incidence of severe neonatal hyperbilirubinemia.

ELIGIBILITY:
Inclusion Criteria:

Term or late-preterm newborn infants with GAs of ≥35 weeks and birth weights of ≥2,000 g were included.

Exclusion Criteria:

All sick newborn infants who were admitted to the intensive care unit.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Term or late-preterm newborn infants from Seventeen hospitals in China were recruited.
Sampling Method: Probability Sample
Enrollment: 13157 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The incidence of severe neonatal hyperbilirubinemia | At the 28 days after birth
  Significant hyperbilirubinemia was defined as any TSB level that exceeded the hour-specific threshold value for phototherapy, according to the guidelines presented by the American Academy of Pediatrics.

SECONDARY OUTCOMES:
Number of participants with risk factors associated with severe neonatal hyperbilirubinemia | At the 28 days after birth
  The risk factors recognized to be associated with significant hyperbilirubinemia in newborns have included gestational age, weight for Gestational Age, delivery mode, gender, previous infant had phototherapy, bruising/cephalahematoma, feeding mode, excessive body weight loss, and early discharge, et al.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Chen, PhD, Study Director — Children's Hospital of Fudan University; Shuping Han, PhD, Study Director — Nanjing Maternity and Child Health Care Hospital; Zhangbin Yu, PhD, Principal Investigator — Nanjing Maternity and Child Health Care Hospital; Chunming Jiang, PhD, Principal Investigator — First Affiliated Hospital of Harbin Medical University; Yan Gao, PhD, Principal Investigator — Jinlin Provincial Maternal and Child Health Hospital; Xiaomei Tong, PhD, Principal Investigator — Peking University Third Hospital; Meihua Pu, PhD, Principal Investigator — Peking University Third Hospital; Hongyun Wang, PhD, Principal Investigator — Inner Mongolia Maternal and Child Health Care Hospital; Kezhan Liu, PhD, Principal Investigator — Shanxi Provincial Maternity and Children's Hospital; Jin Wang, PhD, Principal Investigator — Children's Hospital of Fudan University; Jimei Wang, PhD, Principal Investigator — Obstetrics & Gynecology Hospital of Fudan University; Xiuyong Cheng, PhD, Principal Investigator — The First Affiliated Hospital of Zhengzhou University; Jie Yang, PhD, Principal Investigator — Guangdong Women and Children Hospital; Qiufen Wei, PhD, Principal Investigator — Guangxi Maternal and Child Health Hospital; Zhankui Li, PhD, Principal Investigator — Shanxi Provincial Maternity and Children's Hospital; Mingxia Li, PhD, Principal Investigator — First Affiliated Hospital of Xinjiang Medical University; Changhui Chen, PhD, Principal Investigator — Sichuan Provincial People's Hospital; Ling Liu, PhD, Principal Investigator — Guiyang Maternity and Child Health Care Hospital; Xiaofan Sun, MD, Principal Investigator — Nanjing Maternity and Child Health Care Hospital
Locations (14):
- China (14):
  - Guangdong Maternal and Children's Hospital, Guangzhou Medical College, Guangzhou, Guangdong
  - Guangxi Maternal and Child Health Hospital, Liuchow, Guangxi
  - Guiyang Maternal and Child Health Hospital, Guiyang, Guizhou
  - The First Hospital of Harbin Medical University, Harbin, Heilongjiang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Inner Mongolia Maternal and Child Health Care Hospital, Hohhot, Inner Mongolia
  - Nanjing Maternity and Child Health Care Hospital of Nanjing Medical University, Nanjing, Jiangsu
  - Jinlin Provincial Maternal and Child Health Hospital, Changchun, Jilin
  - Shaanxi Provincial Maternal and Child Health Hospital, Taiyuan, Shaanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The First Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Third Hospital of Peking University, Beijing
  - Gynecology and Obstetrics Hospital, Fudan University, Shanghai
  - Children's Hospital of Fudan University, Shanghai